CLINICAL TRIAL: NCT06700148
Title: A Randomized, Blinded, Peer-controlled Clinical Trial to Evaluate the Safety and Immunogenicity of ACYW135 Group Meningococcal Polysaccharide Conjugate Vaccine (CRM197 Vector) in 7-17 Year Olds
Brief Title: A Clinical Trial of ACYW135 Group Meningococcal Polysaccharide Conjugate Vaccine (CRM197 Vector) in 7 to 17 Year Olds
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: CanSino Biologics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CTP-MCVF-010
Record Dates: First submitted 2024-11-19; First posted 2024-11-21 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2024-11

CONDITIONS: Meningococcal Meningitis
Keywords: Vaccine; Peer controlled; Immunogenicity; Safety; 7-17 years
MeSH Terms: conditions — Meningitis, Meningococcal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACYW135 Group Meningococcal Polysaccharide Conjugate Vaccine (CRM197)(MCV4) (Experimental)
  Interventions: Biological: MCV4
- ACYW135 Group Meningococcal Polysaccharide Vaccine (MPSV4) (Active Comparator)
  Interventions: Biological: MPSV4

INTERVENTIONS:
Biological: MCV4 — 1 dose of MCV4 on Day 0
  Arms: ACYW135 Group Meningococcal Polysaccharide Conjugate Vaccine (CRM197)(MCV4)
Biological: MPSV4 — 1 dose of MPSV4 on Day0
  Arms: ACYW135 Group Meningococcal Polysaccharide Vaccine (MPSV4)

SUMMARY:
This is a randomized, blinded, peer-controlled study. There will be 2 treatment groups, screened subjects were given study numbers in the order of enrollment and randomly assigned to the test and control groups in a 1:1 ratio. Subjects were required to complete a 1-dose immunization program with 0.5 ml of vaccine in both the test and control groups, afterwards some subjects entered the immune persistence group.

ELIGIBILITY:
Inclusion Criteria:

* 7~17 years old at the time of screening
* Volunteers and their legal guardians or delegates have given informed consent, have voluntarily signed an informed consent form, are able and willing to comply with the requirements of the clinical trial protocol, and are able to complete 180 days of study follow-up
* Willingness to discuss medical history with the investigator or physician and to allow access to all medical records related to this trial

Exclusion Criteria:

* Fever on the day of vaccination, axillary temperature >37.0°C
* Have a moderate or severe acute illness/infection
* Positive urine pregnancy test for females of childbearing age, or plan to become pregnant within 30 days after vaccination
* Current meningitis or history of meningitis
* Allergy to certain components or excipients of the drugs used in this clinical trial (mainly including: group A meningococcal podoplanoside, group C meningococcal podoplanoside, group Y meningococcal podoplanoside, group W135 meningococcal podoplanoside, sucrose, mannitol, sodium chloride, dipotassium hydrogen phosphate trihydrate, potassium dihydrogen phosphate)
* History of epilepsy, convulsions or seizures or history or family history of psychiatric disorders
* Previous severe allergic reactions due to drugs or vaccines
* Bleeding constitution or condition associated with prolonged bleeding, which in the opinion of the investigator makes intramuscular injection contraindicated
* Any meningococcal vaccine in the last 1 year
* Any other vaccine within 14 days
* Participation in other studies involving interventional studies within 28 days (<28 days) prior to study entry and/or during study participation
* Other conditions that, in the judgment of the investigator, make participation in this clinical trial unsuitable

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 840 (Actual)
Dates: Start 2024-12-14 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Meningococcal Antibody Positive Conversion Rates and GMT for Groups A, C, Y, and W135 in All Subjects | 30 Days After Immunization
Geometric Mean Titer (GMT) for Groups A, C, Y, and W135 in All Subjects | 30 Days after immunization
Incidence of adverse reactions in all subjects | Within 30 mins after immunization
Incidence of adverse reactions/events in all subjects | Within 7 days after immunization
Incidence of adverse reactions/events in all subjects | Within 30 days after immunization

SECONDARY OUTCOMES:
Meningococcal antibody positivity for groups A, C, Y, and W135 | 30 days after immunization
Geometric mean multiplicity of increase (GMI) for groups A, C, Y, and W135 | 30 days after immunization
Antibody titer ≥1:128 ratio for groups A, C, Y, and W135 | 30 days after immunization
Meningococcal Antibody Positivity for Groups A, C, Y, and W135 in Selected Subjects | 180 days after immunization
GMT for Groups A, C, Y, and W135 in Selected Subjects | 180 days after immunization
GMI for Groups A, C, Y, and W135 in Selected Subjects | 180 days after immunization
Antibody Titer ≥1:128 Ratio for Groups A, C, Y, and W135 in Selected Subjects | 180 days after immunization
Incidence of Serious Adverse Events (SAEs) for all subjects | Within 180 days after immunization

CONTACTS AND LOCATIONS:
Overall Officials: Zhiqiang Xie, Principal Investigator — Henan Center for Disease Control and Prevention
Locations (2):
- China (2):
  - Dengfeng Center for Disease Control and Prevention, Dengfeng
  - Kaifeng Center for Disease Control and Prevention, Kaifeng